CLINICAL TRIAL: NCT04336098
Title: A Phase 1 Study of SRF617 in Patients With Advanced Solid Tumors
Brief Title: Study of SRF617 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Coherus Oncology, Inc. (Industry)
Collaborators: Surface Oncology (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SRF617-101; KEYNOTE-A62 (Other: Merck Sharp & Dohme LLC); MK-3475-A62 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2020-03-30; First posted 2020-04-07 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumor
Keywords: metastatic solid tumors; advanced solid tumors; Phase 1; SRF617; CD39; safety; efficacy; immunotherapy; adenosine pathway; cancer; immuno-oncology; pancreatic cancer; gastric cancer; pembrolizumab; Keytruda®; gemcitabine; albumin-bound paclitaxel; Abraxane®; nab-paclitaxel; gastroesophageal junction adenocarcinoma; GEJ; PD-1; NSCLC; lung cancer
MeSH Terms: conditions — Neoplasms; Pancreatic Neoplasms; Stomach Neoplasms; Lung Neoplasms | interventions — Gemcitabine; Albumin-Bound Paclitaxel; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Monotherapy Dose Escalation (Experimental): The monotherapy dose escalation portion of the study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary efficacy of SRF617 as monotherapy in up to 36 patients with advanced solid tumors.
  Interventions: Drug: SRF617
- Monotherapy Tumor Biopsy Expansion (Experimental): The monotherapy tumor biopsy expansion portion of the study will further evaluate the safety and intratumoral pharmacodynamics of SRF617 monotherapy in up to 20 patients at cleared and recommended phase 2 dose levels.
  Interventions: Drug: SRF617
- Combination Therapy - SRF617 with Gemcitabine + Albumin-bound Paclitaxel Dose Escalation (Experimental): This portion of the study will evaluate the safety, tolerability, PK, and preliminary efficacy of SRF617 in combination with gemcitabine + albumin-bound paclitaxel in patients with locally advanced or metastatic solid tumors.
  Interventions: Drug: SRF617; Drug: Gemcitabine; Drug: Albumin-Bound Paclitaxel
- Combination Therapy - SRF617 with Pembrolizumab Dose Escalation (Experimental): This portion of the study will evaluate the safety, tolerability, PK, and preliminary efficacy of SRF617 in combination with pembrolizumab (Keytruda®) in patients with locally advanced or metastatic solid tumors.
  Interventions: Drug: SRF617; Drug: Pembrolizumab
- Combination Therapy - SRF617 with Gemcitabine + Albumin-bound Paclitaxel Dose Expansion (Experimental): Enrollment at the recommended phase 2 combination dose may be expanded to include approximately 10 additional patients with advanced pancreatic ductal adenocarcinoma (PDAC) to further evaluate safety with SRF617 and gemcitabine + albumin-bound paclitaxel combination therapy.
  Interventions: Drug: SRF617; Drug: Gemcitabine; Drug: Albumin-Bound Paclitaxel
- Combination Therapy - SRF617 with Pembrolizumab Dose Expansion GC/GEJ (Experimental): Enrollment at the recommended phase 2 combination dose may be expanded to include approximately 28 additional patients with 2 anti-PD-(L) 1 naive HER2 negative gastric cancer (GC) or gastroesophageal junction (GEJ) adenocarcinoma to further evaluate safety with SRF617 and pembrolizumab combination therapy.
  Interventions: Drug: SRF617; Drug: Pembrolizumab
- SRF617 + Pembrolizumab + Gemcitabine + Albumin-bound Paclitaxel Quadruplet Dose Expansion (Experimental): Enrollment at the recommended phase 2 combination dose established in the combination dose escalation arms (if recommended phase 2 combination doses differ, the lower of the starting 2 doses will be used) may be expanded to include up to approximately 30 additional patients with advanced 1L PDAC.
  Interventions: Drug: SRF617; Drug: Gemcitabine; Drug: Albumin-Bound Paclitaxel; Drug: Pembrolizumab
- Combination Therapy - SRF617 with Pembrolizumab Dose Expansion anti-PD-L1 GC/GEJ, PD-L1+ NSCLC (Experimental): Enrollment at the recommended phase 2 combination dose may be expanded to include approximately 29 additional patients with anti-PD-(L) 1 relapsed/refractory PD-L1+ HER2 negative gastric cancer (GC) or gastroesophageal junction (GEJ) adenocarcinoma or advanced PD-L1+ NSCLC to further evaluate safety with SRF617 and pembrolizumab combination therapy.
  Interventions: Drug: SRF617; Drug: Pembrolizumab

INTERVENTIONS:
Drug: SRF617 — SRF617 prevents CD39 mediated conversion of adenosine triphosphate (ATP) and adenosine diphosphate (ADP) to adenosine monophosphate (AMP) and phosphate, leading to an increase in extracellular ATP and a reduction in adenosine levels within the tumor microenvironment (TME). There is an important role for extracellular ATP and adenosine in cancer maintenance and progression, and maintaining high levels of ATP (and low levels of adenosine) in the TME may have anticancer therapeutic activity.
Drug: Gemcitabine — Gemcitabine as an intravenous (IV) infusion
  Other Names: Gemzar®
  Arms: Combination Therapy - SRF617 with Gemcitabine + Albumin-bound Paclitaxel Dose Escalation; Combination Therapy - SRF617 with Gemcitabine + Albumin-bound Paclitaxel Dose Expansion; SRF617 + Pembrolizumab + Gemcitabine + Albumin-bound Paclitaxel Quadruplet Dose Expansion
Drug: Albumin-Bound Paclitaxel — Albumin-bound paclitaxel as an IV infusion
  Other Names: Abraxane®
  Arms: Combination Therapy - SRF617 with Gemcitabine + Albumin-bound Paclitaxel Dose Escalation; Combination Therapy - SRF617 with Gemcitabine + Albumin-bound Paclitaxel Dose Expansion; SRF617 + Pembrolizumab + Gemcitabine + Albumin-bound Paclitaxel Quadruplet Dose Expansion
Drug: Pembrolizumab — Pembrolizumab as an IV infusion .
  Other Names: Keytruda®
  Arms: Combination Therapy - SRF617 with Pembrolizumab Dose Escalation; Combination Therapy - SRF617 with Pembrolizumab Dose Expansion GC/GEJ; Combination Therapy - SRF617 with Pembrolizumab Dose Expansion anti-PD-L1 GC/GEJ, PD-L1+ NSCLC; SRF617 + Pembrolizumab + Gemcitabine + Albumin-bound Paclitaxel Quadruplet Dose Expansion

SUMMARY:
A Phase 1, first-in-human, monotherapy and combination dose escalation and expansion study of SRF617.

DETAILED DESCRIPTION:
A Phase 1, open-label, first-in-human, study of SRF617, consisting of a monotherapy dose escalation, a monotherapy tumor biopsy expansion, combination dose escalations, and combination safety and efficacy expansions that will enroll patients with advanced solid tumors. The monotherapy dose escalation portion of the study will evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of SRF617 as monotherapy in patients with advanced solid tumors. The monotherapy tumor biopsy expansion portion of the study will further evaluate the safety and intratumoral pharmacodynamics of SRF617 monotherapy. The combination therapy dose escalation portion of the study will evaluate the safety, tolerability, PK, and preliminary efficacy of SRF617 in combination with gemcitabine + albumin-bound paclitaxel, or SRF617 in combination with pembrolizumab, in patients with locally advanced or metastatic solid tumors. Once the SRF617 combination recommended Phase 2 doses are established, additional patients with select solid tumors may be enrolled in the respective combination expansion arm of the study. An additional quadruplet combination will also be explored in patients with advanced first line (1L) PDAC (i.e., SRF617 + pembrolizumab + gemcitabine + albumin-bound paclitaxel).

ELIGIBILITY:
Abbreviated Inclusion Criteria:

1. Be ≥ 18 years of age on day of signing the informed consent
2. Experienced disease progression during or after standard therapy or were intolerant of standard therapy, and for whom no appropriate therapies are available (based on the judgment of the Investigator). (Exception: PDAC patients in 1L combination expansion arms.)
3. Histological or cytological evidence of advanced, relapsed, or refractory solid tumor cancer that is not a candidate for curative therapy
4. For all patients in the combination expansion arms, have at least 1 lesion that is measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by local site Investigator/radiology. The measurable lesion must be outside of a radiation field if the participant received prior radiation. Lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions.
5. Have tumor tissue that is accessible for pretreatment and on treatment biopsy in the opinion of the Investigator and be willing to undergo pretreatment and on-treatment biopsies per protocol (for patients in the monotherapy tumor biopsy expansion arm only).
6. Adequate renal function
7. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) (≤ 3 x ULN if elevated because of Gilbert's syndrome); patients to be treated with SRF617 in combination with albumin-bound paclitaxel must have total bilirubin ≤ 1.5 × ULN)
8. Aspartate aminotransferase and alanine aminotransferase < 2.5 x ULN (< 5 x ULN if liver metastasis is present)
9. Adequate hematologic function, defined as absolute neutrophil count (ANC) ≥ 1.0 x 109/L, hemoglobin ≥ 8.0 g/dL, and platelet count ≥ 75 x 109/L. Blood cell transfusion to meet enrollment criteria is not allowed
10. Prothrombin time (PT) or international normalized ratio (INR) and activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless the patient is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
11. Eastern Cooperative Oncology Group performance status of 0 to 1
12. For the SRF617 + gemcitabine + albumin-bound paclitaxel expansion arm and SRF617 + pembrolizumab + gemcitabine + albumin-bound paclitaxel quadruplet expansion arm enrolling patients with 1L PDAC only:

    1. Patients with confirmed advanced PDAC naive to any prior systemic treatment
    2. Prior neoadjuvant or adjuvant therapy for PDAC is permitted if neoadjuvant or adjuvant therapy was completed at least 6 months prior to study enrollment. Prior pembrolizumab treatment is not allowed if patient is enrolling in the quadruplet expansion arm.
    3. Patients initially diagnosed with locally advanced PDAC who have undergone chemotherapy then resection and had no evidence of disease are eligible if relapsed or metastatic disease has occurred and if the last dose of chemotherapy was received more than 6 months before study entry
13. For the anti-PD-(L) 1 naïve SRF617+ pembrolizumab combination expansion arm only:

    1. Patients with unresectable locally advanced or metastatic HER2 GEJ who have received a maximum of 2 prior lines of anticancer therapy
    2. Patients must be anti PD(L)-1 treatment naïve
14. For the anti-PD-(L) 1 relapsed/refractor SRF617 + pembrolizumab expansion arm only:

    1. Patients with unresectable locally advanced or metastatic HER2- GC or GEJ adenocarcinoma or unresectable advanced or metastatic NSCLC whose disease is PD-L1+ (defined as CPS ≥ 1 or TPS ≥ 1%).
    2. Must have received at least 1 prior line of systemic anticancer therapy and no more than 4 prior lines of systemic anticancer therapy
    3. Must have anti-PD-(L) 1 relapsed/refractory diseased defined as having progressed on treatment and with anti-PD-(L)1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other immune checkpoint inhibitors or other therapies.
15. Willingness of male and female patients who are not surgically sterile or postmenopausal to use medically acceptable methods of birth control for the duration of the study treatment period (or beginning 14 days before the initiation of pembrolizumab for oral contraception), including 30 days after the last dose of SRF617, or 120 days after the last dose of pembrolizumab for patients in the pembrolizumab combination arms; male patients must refrain from donating sperm during this period. Sexually active men, and women using oral contraceptive pills, should also use barrier contraception with spermicide. Azoospermic male patients and women of child-bearing potential (WCBP) who are continuously not heterosexually active are exempt from contraceptive requirements; however, female patients must still undergo pregnancy testing as described in this section.

Abbreviated Exclusion Criteria:

1. Previously received an anti-CD39 antibody or anti-CD39 targeted therapy. In combination expansion arms, patients cannot have previously received agents that inhibit CD73, A2AR, or A2BR.
2. History of Grade 3 allergic or anaphylactic reaction to any monoclonal antibody therapy (mAb), or any excipient in the study drugs
3. Major surgery within 4 weeks before Screening
4. Unstable or severe uncontrolled medical condition (eg, unstable cardiac function, unstable pulmonary condition including pneumonitis and/or interstitial lung disease, uncontrolled diabetes) or any important medical illness or abnormal laboratory finding that would, in the Investigator's judgment, increase the risk to the patient associated with his or her participation in the study
5. For patients in the anti-PD-(L) 1 naïve SRF617 + pembrolizumab combination expansion arm only:

   1. Discontinuation from previous therapy with an anti programmed cell death ligand 2 (PD-L2) agent or with an agent directed to another stimulatory or co inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX 40, CD137) due to a ≥ Grade 3 immune-related AE
   2. Prior therapy with anti-PD-1 or anti-PD-L1 agents is not permitted
6. Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 21 days before the first dose of study drug Note: Patients who have entered the follow-up phase of an investigational study may participate if it has been at least 21 days after the last dose of the previous investigational agent
7. Received prior radiotherapy within 2 weeks of start of study treatment. Patients must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (≤ 2 weeks of radiotherapy) to non-central nervous system disease.
8. Has received radiation therapy to the lung that is >30Gy within 6 months of the first dose of study treatment
9. Current pneumonitis or history of (non-infectious) pneumonitis requiring steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity of SRF617 | Assessed during first 28 days of treatment
  Evaluation of dose-limiting toxicity (DLT).

SECONDARY OUTCOMES:
Safety Analysis: Summary of adverse events (AEs) and based on treatment-emergent AEs (TEAEs) | Up to 24 months
  Safety and tolerability of SRF617 monotherapy and combination therapy will be assessed by summarizing adverse events (AEs) and will be based on treatment-emergent AEs (TEAEs). A TEAE is an AE that emerges or worsens in the period from the first dose of study drug to 30 days after the last dose of study drug assessed by per CTCAE version 5.0 or higher.
Pharmacokinetics (PK) of SRF617 | Up to 24 months
  Serum concentrations of SRF617 will be collected and analyzed to evaluate the PK of SRF617.
Pharmacodynamics of SRF617 | Up to 24 months
  Pharmacodynamics of SRF617 will be evaluated via serum target occupancy.
Objective response rate (ORR) | Up to 24 months
  ORR will be estimated by the percentage of patients achieving a best overall response of CR or PR per iRECIST.
Duration of response (DoR) | Up to 24 months
  DoR is defined as the time from the first documented response (CR or PR) to documented disease progression as determined by applicable disease criteria, or documented death due to any cause, whichever occurs first.
Disease control rate (DCR) | Up to 24 months
  DCR is defined as the percentage of patients with CR, partial PR, or stable disease lasting a minimum of 12 weeks.
Progression-free survival (PFS) | Up to 24 months
  PFS is defined as the time from the first treatment on study with study drug to documented disease progression as determined by applicable disease criteria or death.
Landmark PFS rate | Up to 24 months
  Landmark PFS is defined as the percentage of patients who have not developed PFS events (ie, death or documented disease progression as determined by applicable disease criteria) at 6 months, 1 year, 1.5 years, and 2 years.
Effect of SRF617 on intratumoral CD39 enzymatic activity | Up to 24 months
  Levels of intratumoral CD39 enzymatic activity will be evaluated in patients receiving pretreatment and on-treatment tumor biopsies via an in situ ATPase histochemistry assay.

CONTACTS AND LOCATIONS:
Overall Officials: Alison O'Neill, MD, Study Chair — Surface Oncology
Locations (10):
- United States (8):
  - City of Hope, Duarte, California
  - The Angeles Clinic and Research Institute, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Mary Crowley Cancer Research, Dallas, Texas
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
- Canada (2):
  - University Health Network-Princess Margaret Cancer Centre, Toronto, Ontario
  - Universite de Montreal - Centre Hospitalier de l'Universite de Montreal (CHUM) - Hopital Notre-Dame, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No